CLINICAL TRIAL: NCT06582108
Title: UNDERSTANDING the RAREST GYNECOLOGICAL CANCERS: a MULTI -OMICS PLATFORM for IMPROVED PATIENTS MANAGEMENT
Acronym: ROAR
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, SCAMBIA GIOVANNI, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: ID 6868
Record Dates: First submitted 2024-08-27; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Uterine Sarcoma; Vulvar Cancer; Non Epithelial Ovarian Cancers (NEOC)
MeSH Terms: conditions — Vulvar Neoplasms | interventions — DNA; RNA; Circulating Tumor DNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Genetic: DNA, RNA, ctDNA, metabolomics — The use of specific assays or global molecular profiling to identify novel biomarkers based on DNA, RNA, protein, lipids, or metabolites obtained from tumor tissue or body fluids

SUMMARY:
Rare gynecological cancers including uterine sarcomas, vulvar and non-epithelial ovarian cancers, are under-studied diseases and the absence of standardized diagnostic and therapeutic approaches or tailored clinical guidelines led to low survival rates and/or poor quality of life outcomes.

The ROAR project aims at increasing the molecular understanding of these diseases in a multidisciplinary, interinstitutional setting including gynecologic oncologists, medical oncologists, phase I researchers, pathologists, molecular pathologist, research nurses, genetists, bioinformatics, psychologists and patients' advocacy groups.

The project will pursue this aim through the following activities:

1. Harmonizing procedures and enabling safe and easy data sharing across all involved institutions; this will be achieved by reviewing the available clinical and molecular data (WP1), establishing an interinstitutional second-opinion board (WP2/Task1), developing a dedicated electronic customized research form (WP2/Task2) and deploying a genomics platform (WP2/Task3).
2. Performing comprehensive somatic and transcriptional profiling as well as immunological landscape assessments on high quality annotated samples stored in a biobank dedicated to rare gynecological cancers; this will require systematic and standardized clinical data and biological samples collection (WP3/WP4), standardization of pre-analytical and sequencing procedures (WP5/6). The board will tailor indications and modalities for genomics and liquid biopsy assessments based on clinical features.
3. Evaluating the clinical impact of the board on rare gynecological cancers management and, through the evidence gathered, implementing diagnostic and therapeutic strategies; this will include analyzing the activities of the board (WP7/Task 1.1), integrating -omics data in the board report (WP7/Task 1.2), evaluating liquid biopsy role in identifying minimal residual disease post-surgery, disease monitoring over time, capability of capturing tumor heterogeneity at baseline and identifying hot spot actionable molecular alterations. Finally, the evidence gathered from the ROAR project, will allow update of clinical guidelines or provide new recommendations for each rare gynecological cancer included. The results of ROAR will also be disseminated through direct access to the integrated platform developed.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old

Histological diagnosis of:

Non-epithelial ovarian tumors Uterine sarcomas Vulvar cancer

Exclusion Criteria:

* Active HIV, HBV, or HCV infection Synchronous neoplasms Non-rare histologies of gynecological malignancies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients with non-epithelial ovarian tumors, 40 with uterine sarcomas, and 120 with vulvar tumors
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To revise available data on RGCs, implement standards of care procedures for RGCs across all involved centers and establish the infrastructure to run the project. | 6 months
Integration and implementation of high quality annotated samples storage, clinical data collection and multi-omics molecular data generation in a data-biobank dedicated to RGCs. | 12 months
Impact of molecular data on clinical management of rare gynecological cancers patients. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No